CLINICAL TRIAL: NCT02382692
Title: Auftreten Von Okkultem Asymptomatischem Liqourverlust Nach Nebenhöhlenoperationen Eine Prospektive Kohortenstudie
Brief Title: Cerebrospinal Fluid Rhinorrhea After Functional Endoscopic Sinus Surgery
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SM_27_02_2015
Record Dates: First submitted 2015-03-02; First posted 2015-03-09 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cerebrospinal Fluid Leakage
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA Samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Sinus surgery is a common procedure. A potential complication is injuring the membranes of the brain. This can lead to leakage of brain fluid through the nose. We would like to estimate the incident rates of that complication. At the end of the operation, a thin gauze is inserted into the nose on both sides in addition to the usual tampon. This gauze will be analyzed at the laboratory for beta-2-transferrin, which is a biomarker for brain liquid.

DETAILED DESCRIPTION:
Sinus surgery is a common procedure in rhinology for the treatment of chronic inflammation, tumors and other pathologies. These procedures are performed in the immediate vicinity of the skull base. The risk of injuring the membranes covering the brain in a way that requires further treatment is less than 1% [ 1]. Such Injuries to the skull base could lead to the loss of cerebrospinal fluid (CSF). The destruction of the natural barrier raises the potential risk of ascending infections of the membranes and the brain itself from the nose. Leakage of cerebrospinal fluid in the usually bloody surgical field of view is not always distinguishable and is sometimes only noticed postoperatively. The spontaneous closure of a leaky membrane of the brain without further surgical treatment is known. This is why small traumata in the skull base often remain undetected.

At the end of the operation, a thin gauze is inserted into the nose on both sides in addition to the usual tampon. The tampon and the additional gauze are removed the day after the operation and will be sent with a tube of venous blood to the laboratory. The gauze and the venous blood will be checked for beta-2-transferrin, which is a biomarker for cerebrospinal fluid.

During further clinical standard controls will the patient be asked about symptoms of fluid leak through the nose.

If positive, regardless to this study, the patient must have an additional CT scan of the sinuses and another blood sample checking for beta-2-transferrin.

ELIGIBILITY:
Inclusion Criteria:

* All patients with planned sinus surgery in terms of Ethmoidektomie / Sphenoethmoidektomie or Frontosphenoethmoidektomie
* Male and female patients aged 18 to 99 years
* Written consent of the participating person after the enlightenment

Exclusion Criteria:

* Olanned or accidental opening of the skull base
* Tumor in the skull base
* Pre-existing known rhinoliquorrhoe
* Lack of understanding the study or investigation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication to a sinus intervention without planned opening of the skull base
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Beta-2-Transferrin positive or negative | 1 day postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soyka MB, Holzmann D. Correlation of complications during endoscopic sinus surgery with surgeon skill level and extent of surgery. Am J Rhinol. 2005 May-Jun;19(3):274-81. PMID 16011134